CLINICAL TRIAL: NCT05346692
Title: A Prospective, Double-Arm Pilot Study to Investigate the Safety, Feasibility and Acceptability of a Digital Mindfulness Intervention Following Open Abdominal Surgery for Cancer
Brief Title: Digital Meditation for Postoperative Pain Control After Abdominal Surgery for Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Viraj Master, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003299; EU5450-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-03-28; First posted 2022-04-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Pain Survey) (Active Comparator): Patients complete pain survey via text message daily for 10 days after surgery. Patients also complete telephone interview 2 weeks after surgery.
  Interventions: Other: Survey Administration; Other: Interview
- Arm 2 (Mindfulness Intervention) (Experimental): Patients complete mindfulness intervention via text message daily for 10 days after surgery. Patients also complete telephone interview 2 weeks after surgery.
  Interventions: Other: Text Message-Based Navigation Intervention; Other: Interview

INTERVENTIONS:
Other: Survey Administration — Complete Survey
  Arms: Arm I (Pain Survey)
Other: Interview — Complete Interview
  Arms: Arm I (Pain Survey)
Other: Text Message-Based Navigation Intervention — Complete mindfulness intervention
  Other Names: Automated Text Message-Based Navigation, Text Message-Based Navigation
  Arms: Arm 2 (Mindfulness Intervention)
Other: Interview — Complete interview
  Arms: Arm 2 (Mindfulness Intervention)

SUMMARY:
This phase I trial tests a digital meditation for postoperative pain control after abdominal surgery for cancer. Mindfulness interventions such as guided meditation may improve pain control and decrease stress. Including a brief mindfulness intervention administered via test messages as part of postoperative care may improve pain severity, decrease opioid use, and improve patient responses to non-surgical treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate and define anticipated and unanticipated adverse events (AEs) related to a daily virtual mindfulness intervention delivered via short message service (SMS) text messaging and to test its safety in the postoperative period amongst patients with cancer.

II. To determine the feasibility and acceptability of a novel, brief mindfulness intervention delivered via SMS text messaging in the postoperative period amongst patients undergoing surgery for cancer.

III. To determine the feasibility and acceptability of an artificial intelligence platform to deliver and receive SMS text messages for the purpose of delivering pain assessment tools and collecting and storing pain-specific and patient reported outcomes.

OUTLINE: Patients are assigned to 1 of 2 arms. ARM I: Patients complete pain survey via text message daily for 10 days after surgery. Patients also complete telephone interview 2 weeks after surgery.

ARM II: Patients complete mindfulness intervention via text message daily for 10 days after surgery. Patients also complete telephone interview 2 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age
* Open abdominal surgery for cancer
* Ownership of smartphone (iOS or Android operating systems) with SMS texting capabilities
* Ability to read
* Ability to understand the purposes and risk of the study and willingly give standard written informed consent for treatment established by each participating institution.

Exclusion Criteria:

* Patients with contraindications to abdominal surgery and/or general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 months
  Adverse events (AEs) will be reported, and summarized using frequencies and percentages. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study intervention. Unexpected AEs will be summarized descriptively. The most common adverse events reported within the mindfulness literature anxiety, depression, and cognitive anomalies. The overall prevalence of meditation adverse events is 8%, which is similar to those reported for psychotherapy practice in general.
Feasibility of intervention and mode of delivery | Up to 12 months
  Feasibility for each arm is defined as completion of at least 50% of the program.The proportion completing at least 50% of the program will be compared to a null proportion of 20% completing at least 50% of the program using a one-sample Z-test.

SECONDARY OUTCOMES:
Intervention and mode of delivery utilizing the Client Satisfaction Survey (CSQ-8) | Up to 12 months
  Acceptability of intervention and mode of delivery will include quantitative and qualitative analyses. Quantitative analysis will include the Client Satisfaction Survey (CSQ-8). The CSQ-8 focuses on participant satisfaction with the intervention received, including:
  1. the overall quality
  2. perception of the program's ability to meet their needs
  3. amount of help received
  4. the extent to which this program helped them deal with recovery after surgery. The CSQ-8 has demonstrated good internal consistency, test-retest reliability, and sensitivity10.
Intervention and mode of delivery utilizing the System Usability Scale (SUS) | Up to 12 months
  Acceptability of intervention and mode of delivery will include quantitative and qualitative analyses. Quantitative analysis will include the System Usability Scale (SUS) administered to all participants at study completion of the study to all participants.
  The SUS is a 10-item scale that examines the perceived usability of a technology and is commonly used in evaluating mobile apps. The SUS has demonstrated good reliability in other studies.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Diller, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No